CLINICAL TRIAL: NCT06209983
Title: The Effect of Enhanced Recovery After Surgery (ERAS) in Gastric Cancer Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201809008RINC
Record Dates: First submitted 2023-10-16; First posted 2024-01-18 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-10

CONDITIONS: Anesthesiology; General Surgery
Keywords: ERAS; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm E (Experimental): 1. Preoperative preparation: shorten the fasting time, take a small amount of sugar water two hours before the surgery, and reduce excessive bowel preparation.
  2. Intraoperative care: multi-model analgesia (mainly epidural analgesia), sleep depth monitoring, warm air blanket to avoid hypothermia.
  3. Postoperative care: focus on pain relief methods (such as oral analgesics, patient-controlled epidural analgesia), early postoperative feeding (try drinking water on the first day after surgery, liquid diet on the second day, and soft diet on the third day), early removal of invasive tubes such as nasogastric tubes, intravenous catheters, and urinary catheters, and medication to prevent postoperative nausea and vomiting.
  Interventions: Procedure: ERAS
- Arm H (Placebo Comparator): 1. Preoperative preparation: overnight fasting preparation, bowel preparation.
  2. Intraoperative care: traditional pain care (intravenous analgesics), sleep depth monitoring, warm air blanket, central venous pressure and body water monitoring indicators, traditional muscle tension relaxation treatment and the use of health insurance antagonist drugs (Neostigmine).
  3. Postoperative care: patient-controlled intravenous drip for postoperative pain relief, oral feeing (rice porridge) on the postoperative day 5, and according to the progression of patient condition, step by step to removal of invasive tubes such as nasogastric tubes, intravenous catheters, and urinary catheters.
  Interventions: Procedure: Conventional care

INTERVENTIONS:
Procedure: ERAS — 1. Preoperative preparation: shorten the fasting time, take a small amount of sugar water two hours before the surgery, and reduce excessive bowel preparation.
  2. Intraoperative care: multi-model analgesia (mainly epidural analgesia), sleep depth monitoring, warm air blanket to avoid hypothermia.
  3. Postoperative care: focus on pain relief methods (such as oral analgesics, patient-controlled epidural analgesia), early postoperative feeding (try drinking water on the first day after surgery, liquid diet on the second day, and soft diet on the third day), early removal of invasive tubes such as nasogastric tubes, intravenous catheters, and urinary catheters, and medication to prevent postoperative nausea and vomiting.
  Arms: Arm E
Procedure: Conventional care — 1. Preoperative preparation: overnight fasting preparation, bowel preparation.
  2. Intraoperative care: traditional pain care (intravenous analgesics), sleep depth monitoring, warm air blanket, central venous pressure and body water monitoring indicators, traditional muscle tension relaxation treatment and the use of health insurance antagonist drugs (Neostigmine).
  3. Postoperative care: patient-controlled intravenous drip for postoperative pain relief, oral feeing (rice porridge) on the postoperative day 5, and according to the progression of patient condition, step by step to removal of invasive tubes such as nasogastric tubes, intravenous catheters, and urinary catheters.
  Arms: Arm H

SUMMARY:
The investigators aimed to clarify the clinical relevance of the ERAS protocol by evaluating the perioperative course in patients undergoing laparoscopic gastric cancer surgery.

DETAILED DESCRIPTION:
Gastric cancer is 7th common malignant disease in Taiwan, accounting for 3000 new cases per year. The main treatment of gastric cancer is radical gastrectomy and lymph nodes dissection, which is associated with 13.0~46 % of surgical morbidities. To minimize the surgical morbidities and enhance patients' recovery, perioperative management is mandatory. Enhanced Recovery After Surgery (ERAS) is a multimodal, multidisciplinary approach to the care of the surgical patient. ERAS process implementation involves a team consisting of surgeons, anesthetists, an ERAS coordinator, and staff from units that care for the surgical patient. The main elements of ERAS include carbohydrate loading before surgery, minimally invasive approaches, balanced management of intravenous fluids, multimodal pain management, early mobilization, and early oral feeding, etc. Some prospective studies have shown its effectiveness in reduce surgical morbidity and hospital stay in colorectal surgery. In Taiwan, there was only limited report to study the use of ERAS in gastric cancer surgery. The investigators would like to integrate these perioperative interventions into the ERAS program, and test its effectiveness in gastric cancer patients undergoing radical gastrectomy at NTUH.

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmed as gastric adenocarcinoma;
* Gastric cancer patients who will undergo subtotal gastrectomy.

Exclusion Criteria:

* Advanced gastric cancer with gastric outlet obstruction;
* Epidural catheter placement contraindicated or inexecutable;
* Have other cancers that have received chemotherapy or radiation therapy;
* Coagulation abnormalities;
* Pregnancy;
* Severe dysfunction of major organs (e.g., heart failure, chronic obstructive pulmonary disease, liver cirrhosis, end-stage renal disease)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2018-12-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | From date of admission until the date of discharge, assessed up to 2 weeks.
  When patient discharge.

SECONDARY OUTCOMES:
Complication rates | 28 days
  The complication rates means if there are any complications occur.

OTHER OUTCOMES:
Readmission rates | within 28 days
  when the patient is readmitted to the hospital
costs of hospitalization | From date of admission until the date of discharge, assessed up to 2 weeks.
  Total medical expenses incurred during the admission period.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No